CLINICAL TRIAL: NCT02688296
Title: The Use Of A Fibular Intramedullary Nail For Fixation For Unstable Fibula Fractures
Brief Title: Effectiveness Of The Fibulock Intramedullary Nail
Acronym: Fibulock
Status: Completed | Type: Observational
Sponsor: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FIB-001
Record Dates: First submitted 2016-02-10; First posted 2016-02-23 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Fibula Fracture
MeSH Terms: conditions — Fibula Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Pilon Fractures: Patients who are implanted with Fibulock and have a Pilon fracture
  Interventions: Device: Fibulock
- High Risk Patients: Patients who are implanted with Fibulock and are at high risk of complications from ankle surgery due to conditions such as diabetes, advanced age or osteoporosis
  Interventions: Device: Fibulock
- Otherwise Healthy Patients: Patients implanted with Fibulock who are healthy other than their ankle fracture
  Interventions: Device: Fibulock

INTERVENTIONS:
Device: Fibulock — Fibulock intramedullary implant will be used to repair fibula fractures

SUMMARY:
The objective of this post-market clinical study is to evaluate efficacy outcomes and complication rates in patients who have received the Fibulock™ Intramedullary Nail.

DETAILED DESCRIPTION:
This is a retrospective/prospective, multi-site observational study, designed to evaluate the clinical outcomes and complication rates in subjects who were previously implanted with a Fibulock™ intramedullary nail.

Patients will be screened for eligibility and subgroupings. Informed consent will be obtained from those who meet screening criteria and are interested in participating in the study.

Sites will be asked to enroll subjects according to past treatment, with the Fibulock™ intramedullary nail for unstable fibula fracture. The sites will enroll subjects in the study based on inclusion/exclusion criteria.

Patient pre-operative, intra-operative and post-operative records will be reviewed retrospectively. Once enrolled, subjects will undergo an evaluation of fracture outcome and complete a VAS pain score, SF-12, and Foot Function Index at 26 weeks and again at 52 weeks post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* An unstable fibula fracture.
* Must be less than 31 weeks post-implantation
* Must have received surgical treatment with the Fibulock Intramedullary Nail for their unstable fibula - fracture
* Male or female greater than or equal to 18 years of age and skeletally mature.
* Able to understand the requirements of the study, provide a written informed consent and comply with the study protocol
* Ability to understand and provide written authorization for use and disclosure of personal health information.

Exclusion Criteria:

* Patients who are not implanted with a Sonoma Fibulock IM Nail

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who received the Fibulock Intramedullary Nailand are at least 12 weeks post implant, but less than 31 weeks post implant.
Sampling Method: Non-Probability Sample
Enrollment: 34 (Actual)
Dates: Start 2016-05-24 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Efficacy Assessment post implantation with Fibulock Intramedullary Nail assessed using lateral and mortice view x-rays | 26 weeks
  Lateral and mortice view x-rays at 26 weeks

SECONDARY OUTCOMES:
Visual Analog Scale | 26 weeks and 52 weeks
  Patient self reported pain intensity.
SF 12 | 26 weeks and 52 weeks
  SF 12 is a Health Survey that uses just 12 questions to measure functional health and well-being from the patient's point of view.
Foot Function Index | 26 weeks and 52 weeks
  The Foot Function Index (FFI) is used to measure the impact of foot pathology on function in terms of pain, disability and activity restriction.

CONTACTS AND LOCATIONS:
Overall Officials: Terrence Philbin, MD, Principal Investigator — Orthopedic Foot & Ankle; Selene Parekh, MD, Principal Investigator — NCOC; Chris Hodgkins, MD, Principal Investigator — Baptist Health South Florida, Inc.
Locations (3):
- United States (3):
  - Baptist Health South Florida, Miami, Florida
  - NCOC, Durham, North Carolina
  - Orthopedic Foot & Ankle Center, Westerville, Ohio

IPD SHARING:
Plan to Share IPD: No